CLINICAL TRIAL: NCT04228146
Title: Parallel Group Randomized Controlled Trial on the Effect of a Smartphone-delivered Cognitive Behavioral Therapy for Insomnia on People With Major Depression and Insomnia
Brief Title: Self-help Smartphone-delivered Cognitive Behavioral Therapy for Insomnia in People With Depression and Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Christian S. Chan, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1810026
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Sleep Initiation and Maintenance Disorders; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I condition (Experimental): Participants in the CBT-I condition start the 6-week CBT-I immediately after randomization, complete the post-intervention assessment right after they finish the treatment, and complete the follow-up assessment six weeks after the post-intervention assessment.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Waitlist control condition (Other): Participants in the waitlist control group complete the post-intervention assessment six weeks after the baseline assessment, start CBT-I (equivalent to that of the CBT-I group) immediately after completing the post-intervention assessment, and complete the follow-up assessment right after they finish the 6-week CBT-I.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Immediate access to the self-help CBT-I treatment, content of which is based on the translated Chinese version of a well-established CBT-I treatment manual entitled "Insomnia: A Clinician's Guide to Assessment and Treatment". CBT-I aims at changing dysfunctional cognitive beliefs and maladaptive behaviors that contribute to the maintenance of insomnia. The self-help CBT-I treatment is delivered in Chinese language in six consecutive weekly modules via a smartphone application known as proACT-S. Duration of each module is around 45 to 60 minutes.
  Arms: CBT-I condition
Other: Waitlist Control — Delay access to the self-help CBT-I treatment.
  Arms: Waitlist control condition

SUMMARY:
This randomized controlled trial aims to examine the effectiveness of a self-help smartphone-delivered cognitive behavioral therapy for insomnia, compared to a waitlist control, in treating people with major depression and insomnia in Hong Kong.

DETAILED DESCRIPTION:
Depression is a major public health concern. Emerging research has shown that cognitive behavioral therapy for insomnia (CBT-I) is effective in treating individuals with comorbid insomnia and depression. Traditional face-to-face CBT-I encounters many obstacles related to feasibility, accessibility, and help-seeking stigma. CBT-I delivered via smartphone application could be a potential solution. This two-arm parallel randomized controlled trial (RCT) aims to examine the effectiveness of a smartphone-based self-help CBT-I with a waitlist control group in treating people with major depression and insomnia in Hong Kong.

Participants complete an online rapid screening, followed by a telephone diagnostic interview. Those who meet the eligibility criteria are randomized in a ratio of 1:1 to receive either CBT-I immediately or to a waitlist control condition. The CBT-I consists of six weekly modules and is delivered through a smartphone application known as proACT-S. An online randomized algorithm is used to perform randomization to ensure allocation concealment. The primary outcomes are changes over the measurement points in sleep quality, insomnia severity and depression severity. The secondary outcomes include changes over the measurement points in anxiety, subjective health, treatment expectancy, and acceptability of treatment. Assessments are administered at baseline, post-intervention, and 6-week follow up. The recruitment is underway. Important adverse events, if any, are documented. Multilevel linear mixed model based on intention-to-treat principle will be conducted to examine the effectiveness of the CBT-I intervention

Participants in the CBT-I condition will start CBT-I immediately after randomization; while participants in the waitlist control group will start CBT-I (equivalent to that of the CBT-I group) immediately after completing the post-intervention assessment. It is hypothesized that, after the intervention, participants in the CBT-I condition will report a greater decrease in poor sleep quality, depression severity and insomnia severity than those in the waitlist control condition. It is also hypothesized that the reduction in poor sleep quality, depression severity and insomnia severity observed in the CBT-I condition will be maintained at 6-week follow-up. Furthermore, it is hypothesized that participants in the waitlist control condition will report a significant decrease in poor sleep quality, depression severity and insomnia severity after receiving CBT-I.

ELIGIBILITY:
Stage 1 Screening (Online Survey) Inclusion Criteria:

* Hong Kong residents
* age ≥ 18 years
* predominant complaint of difficulty initiating or maintaining sleep or early morning awakening or non-restorative sleep with associated distress or impairment in social, occupational and other important areas of functioning for at least three nights per week for at least three months
* Insomnia Severity Index score ≥ 8
* Patient Health Questionnaire (PHQ-9) score ≥ 10
* being able to read Chinese and type Chinese or English
* have a smartphone device (iOS or Android operating system) with Internet access
* have a regular email address
* willing to give informed consent and comply with the trial protocol

Stage 1 Screening (Online Survey) Exclusion Criteria:

* Beck Depression Inventory II (BDI-II) suicidal ideation score ≥ 2
* receiving concurrent psychological treatment at least once per month
* former proACT-S pilot clinical trial participants
* currently taking prescribed psychiatric drugs such as antidepressants, tranquilizers, sleeping pills regularly
* carrying a diagnosis of psychosis or schizophrenia
* participating in any other academic studies or clinical trials related to insomnia and/or depression

Stage 2 Screening (Telephone Diagnostic Interview) Inclusion Criteria

* difficulty initiating sleep, maintaining sleep, or early-morning awakening with inability to return to sleep at least once in the past two weeks
* International Statistical Classification of Diseases and Related Health Problems - Tenth Revision diagnosis of depression (F32.00, F32.01, F32.10, F32.11, F32.2)

Stage 2 Screening (Telephone Diagnostic Interview) Exclusion Criteria

* having concurrent psychological treatment at least once per month
* currently taking prescribed psychiatric drugs such as antidepressants, tranquilizers, sleeping pills regularly
* carrying a diagnosis of psychosis or schizophrenia
* participating in any other academic studies or clinical trials related to insomnia and/or depression
* having current suicidal plans or acts or have had suicidal plans or acts within the past 12 months

Main Study Trial Withdrawal Criteria

* have concurrent psychological treatment at least once per month
* are taking prescribed psychiatric drugs such as antidepressants, tranquilizers, sleeping pills regularly
* are being diagnosed with psychosis or schizophrenia
* are participating in any other academic studies or clinical trials related to insomnia and/or depression
* have suicidal ideations defined as scoring ≥ 2 on the BDI-II suicidal ideation item
* have experienced serious diseases, significant life events, hospitalization, or fatalities
* withdraw their consent
* do not complete each assessment within two weeks, do not submit consent within two weeks after proACT-S personal account registration, or do not log into proACT-S within two weeks after random group assignment. (waitlist control group) fail the cross-condition contamination check

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes over the measurement points in Center for Epidemiologic Studies Depression Scale | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures the severity of depressive symptoms during the past week. Range from 0 to 60, where a higher value indicates more severe depressive symptoms.
Changes over the measurement points in Insomnia Severity Index | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures the severity of insomnia symptoms and the associated daytime impairment over the past two weeks. Range from 0 to 21, where a higher value indicates more severe insomnia symptoms.
Changes over the measurement points in Pittsburgh Sleep Quality Index | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures sleep quality and disturbances during the past month. It has seven components, namely, sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of hypnotics, and daytime dysfunction. Range from 0 to 21, where a higher value indicates poorer sleep quality.

SECONDARY OUTCOMES:
Changes over measurement points in SF-12 Version 1 Physical Scale | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures subjective physical health status during the past four weeks. A higher value indicates better subjective physical health.
Changes over measurement points in SF-12 Version 1 Mental Scale | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures subjective physical health status during the past four weeks. A higher value indicates better subjective mental health.
Changes over measurement points in Hospital Anxiety and Depression Scale - Anxiety subscale | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures severity of anxiety symptoms during the past week. Range from 0 to 21, where a higher value indicates more severe anxiety symptoms.

OTHER OUTCOMES:
Changes over measurement points in Modified Credibility/Expectancy Questionnaire (Credibility Scores) | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures participants' perceived treatment credibility. A higher value indicates higher levels of perceived treatment credibility.
Changes over measurement points in Modified Credibility/Expectancy Questionnaire (Expectancy Scores) | Baseline, post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures participants' perceived treatment expectancy. A higher value indicates higher levels of perceived treatment expectancy.
Modified Participant Acceptability/Usability Rating Scale | Post-intervention: 6 weeks after CBT-I initiation, 6-week follow up
  Measures participants' subjective evaluation of the treatment received via the smartphone application. A higher value indicates higher levels of perceived treatment acceptability.
Demographics | Stage 1 screening (online survey): First day of enrollment
  Measures Participants' age, education level, marital status, occupation, and gender
Clinical comorbidity | Stage 2 screening (telephone diagnostic interview): Up to 3 months after enrollment
  Measures current diagnosis of four major comorbidities (generalized anxiety disorder, phobias, obsessive compulsive disorder, and panic disorder).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, The University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chan CS, Wong CYF, Yu BYM, Hui VKY, Ho FYY, Cuijpers P. Treating depression with a smartphone-delivered self-help cognitive behavioral therapy for insomnia: a parallel-group randomized controlled trial. Psychol Med. 2023 Apr;53(5):1799-1813. doi: 10.1017/S0033291721003421. Epub 2021 Aug 23. PMID 37310329
- [Derived] Hui VK, Wong CY, Ma EK, Ho FY, Chan CS. Treating depression with a smartphone-delivered self-help cognitive behavioral therapy for insomnia: study protocol for a parallel group randomized controlled trial. Trials. 2020 Oct 9;21(1):843. doi: 10.1186/s13063-020-04778-1. PMID 33036655